CLINICAL TRIAL: NCT02258919
Title: Swiss Trial of Decompressive Craniectomy Versus Best Medical Treatment of Spontaneous Supratentorial Intracerebral Hemorrhage (SWITCH): a Randomized Controlled Trial
Brief Title: Decompressive Hemicraniectomy in Intracerebral Hemorrhage
Acronym: SWITCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 163/14; 32003B_150009 (Other Grant/Funding Number: SNF)
Record Dates: First submitted 2014-09-30; First posted 2014-10-08 (Estimated); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Hemorrhage
Keywords: Intracerebral hemorrhage; Decompressive craniectomy; Randomized controlled trial; Acute stroke
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke | interventions — Decompressive Craniectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decompressive craniectomy and best medical treatment (Experimental): Decompressive craniectomy and best medical treatment
  Interventions: Procedure: Decompressive craniectomy (DC) and best medical treatment
- Best medical treatment (Active Comparator): Best medical treatment
  Interventions: Procedure: Best medical treatment

INTERVENTIONS:
Procedure: Decompressive craniectomy (DC) and best medical treatment — Decompressive craniectomy:
  All patients in the treatment group will receive DC of at least 12 cm according to institutional guidelines and a published surgical protocol.
  Best medical treatment:
  Best medical treatment is based on American Heart Association/American Stroke Association (AHA/ASA) and European Stroke Organisation (ESO) as published in the current protocol from 2010 and 2014 respectively.
  Arms: Decompressive craniectomy and best medical treatment
Procedure: Best medical treatment — Best medical treatment is based on American Heart Association/American Stroke Association (AHA/ASA) and European Stroke Organisation (ESO) as published in the current protocol from 2010 and 2014 respectively.
  Arms: Best medical treatment

SUMMARY:
Spontaneous intracerebral hemorrhage (ICH) remains a devastating disease with mortality rates up to 52% at 30 days. It is a major public health problem with an annual incidence of 10-30 per 100'000 population, accounting for 2 million (10-15%) of about 15 million strokes worldwide each year. The strategy of decompressive craniectomy (DC) is beneficial in patients with malignant middle cerebral artery (MCA) infarction. Based on the common pathophysiological mechanisms of these two conditions, this procedure is also frequently performed in patients with ICH, but is has not yet been investigated in a randomized trial.

The primary objective of this randomized controlled trial is to determine whether decompressive surgery and best medical treatment in patients with spontaneous ICH will improve outcome compared to best medical treatment only.

Secondary objectives are to analyze mortality, dependency and quality of life. Safety endpoints are to determine cause of any mortality and the rate of medical and surgical complications after DC compared with best medical treatment alone.

DETAILED DESCRIPTION:
Background

Spontaneous intracerebral hemorrhage (ICH) remains a devastating disease with mortality rates up to 52% at 30 days. It is a major public health problem with an annual incidence of 10-30 per 100'000 population, accounting for 2 million (10-15%) of about 15 million strokes worldwide each year. One-third of patients with ICH die within one month and the majority of survivors remain handicapped. Neurological injury resulting from ICH is mediated by the mass effect of the hematoma, secondary to brain edema and/or both mechanisms. Treatment of ICH is one of the major unresolved issues of acute stroke treatment. The International Surgical Trials in Intracerebral Hemorrhage (STICH and STICH II) and other randomized controlled trials did not show any superiority of surgical treatment compared to conservative treatment approaches. Nevertheless, surgical treatment in ICH remains a matter of debate and attempts to improve outcome using surgical therapy are still ongoing. Many efforts are made to minimize the invasiveness of operative procedures such as clot evacuation. However, direct surgical interventions aiming at the removal of the hematoma have failed to improve neurological outcome for most subtypes of ICH, especially deep-seated hematomas. The trauma of open craniotomy and especially trauma to the brain parenchyma for hematoma evacuation are considered to outweigh the benefits of surgery.

Decompressive craniectomy (DC), which is beneficial in patients with malignant middle cerebral artery (MCA) infarction, may indirectly relieve the mass effect, decrease perihematomal tissue pressure, improve blood flow, reduce secondary brain damage and improve outcome without further damage to the brain due to surgery. Consequently, DC has been established as a standard surgical therapy for patients with malignant MCA infarction with a level of evidence grade 2. Decompressive craniectomy for acute stroke is one of the most effective treatments available: the number needed to be treated to save one patient's life is 2. Decompressive craniectomy is also a standard therapeutic procedure in patients with ICH due to sinus venous thrombosis, herpes encephalitis, or ruptured intracranial aneurysms. In patients with traumatic brain injury DC is a standard therapy to reduce elevated intracranial pressure. The investigators and others assessed whether DC is feasible and beneficial in patients with spontaneous intracranial hemorrhage. The investigators showed in a previous retrospective trial that DC in patients with supratentorial ICH is safe and feasible and may reduce mortality compared to matched controls with best medical treatment alone. The limitations of the feasibility trial are its retrospective design, the small sample size and the inhomogeneity of the patient cohort with respect to the origin of ICH. Furthermore, in the feasibility trial the decision for DC was taken on an individual basis rather than according to a strict protocol, introducing a potential selection bias. Nevertheless, the preliminary results are encouraging. Recently, three human trials, one animal study, one meta-analysis, and one original contribution have been published on this topic. However, no prospective randomized trial has ever assessed whether DC without hematoma evacuation in patients with acute ICH improves outcome. All recent studies showed promising results and all call for the initiation of a randomized controlled trial.

Objective

The primary objective of this randomized controlled trial is to determine whether decompressive surgery and best medical treatment in patients with spontaneous ICH will improve outcome compared to best medical treatment only.

Secondary objectives are to analyze mortality, dependency and quality of life. Safety endpoints are to determine cause of any mortality and the rate of medical and surgical complications after DC compared with best medical treatment alone.

Methods

All patients with a suspected intracerebral hemorrhage will be considered for this trial. Randomization of eligible patients will be performed within 66 hours after ictus in patients with stable clot volume and surgery no later than 6 hours after randomization. Patients randomized to the control group will receive best medical treatment according to international guidelines. Patients randomized to the treatment group will receive best medical treatment and a DC of at least 12cm according to institutional guidelines and a surgical protocol. The primary outcome death and dependency at 6 months will be assessed by a trained person unaware of treatment allocation. Favorable outcome is defined as a modified Rankin Scale (mRS) score of 0 to 4, poor outcome as modified Rankin Scale score of 5 or 6.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient or of patient's next of kin plus consent of an independent physician if patient is unable to consent before randomization
* Acute stroke syndrome due to a spontaneous ICH, defined as the sudden occurrence of bleeding into the parenchyma of the basal ganglia and/or thalamus that may extend into the ventricles and into the cerebral lobes, and into the subarachnoid space, confirmed by clinical history and imaging
* Age: ≥18 to ≤75 years
* Glasgow coma scale (GCS) <14 and >7
* Neurological deficit with a NIHSS score of ≥10 and ≤30
* Able to be randomly assigned to surgical treatment within 66 hours after ictus
* Surgery performed not later than 6 hours after randomization
* Volume of hematoma ≥30 ml and ≤100 ml
* Stable clot volume
* International normalized ratio (INR) <1.5, thrombocytes >100 T/ml

Exclusion Criteria

* ICH due to known or suspected structural abnormality in the brain (e.g., intracranial aneurysm, brain arteriovenous malformation, brain tumor) or brain trauma, or previous stroke thrombolysis
* Cerebellar or brainstem hemorrhage
* Exclusive lobar hemorrhage
* Known advanced dementia or significant pre-stroke disability
* Concomitant medical illness that would interfere with outcome assessment and follow-up
* Randomization not possible within 66 hours after ictus
* Pregnancy
* Prior major brain surgery within <6 month or prior DC
* Foreseeable difficulties in follow-up due to geographic reasons
* Known definite contraindication for a surgical procedure
* A very high likelihood that the patient will die within the next 24 hours on the basis of clinical and/or radiological criteria
* Previous participation in this trial or in another ongoing investigational trial
* Prior symptomatic ICH
* ICH secondary to thrombolysis
* Bilateral areactive pupils

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Score in modified Rankin Scale (mRS) | 6 months
  Assessed by telephone interview

SECONDARY OUTCOMES:
Mortality | 7 days, 30 days, 180 days, 12 months
mRS score of 0-3 versus 4-6 | 30 days, 180 days, 12 months
Categorical shift in mRS score | 180 days, 12 months
Quality of life | 180 days, 12 months
Death and intracranial hemorrhage | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Urs Fischer, Prof. Dr. med., Study Director — Dep. of Neurology, Inselspital Bern; Jürgen Beck, Prof. Dr. med., Study Chair — Dep. of Neurosurgery, Inselspital Bern
Locations (32):
- Universitätsklinik für Neurochirurgie, Kepler Universitätsklinikum Linz, Linz, Austria
- UZ Leuven, Leuven, Belgium
- Department of Neurology, Helsinki University Central Hospital, Helsinki, Finland
- France (2):
  - Centre Hospitalier Universitaire de Caen, Caen
  - Fondation Adolphe de Rothschild, Paris
- Germany (18):
  - Klinik für Neurochirurgie, Universitätsklinikum Schleswig Holstein, Lübeck, Schleswig-Holstein
  - Klinik für Neurochirugie, Helios Klinikum Erfurt, Erfurt, Thuringia
  - Klinik für Neurochirurgie Uniklinik RWTH Aachen, Aachen
  - Department of Neurosurgery, Charité - Universitätsmedizin Berlin, Berlin
  - Klinik und Poliklinik für Neurochirurgie, Universitätsklinikum Bonn, Bonn
  - Klinik für Neurochirurgie, Universitätsklinikum Düsseldorf, Düsseldorf
  - Neurologische Klinik, Universitätsklinikum Erlangen, Erlangen
  - Klinik für Neurochirurgie, Universitätsklinikum Essen (AöR), Essen
  - Zentrum der Neurologie und Neurochirurgie, Universitätsklinikum Frankfurt, Frankfurt
  - Klinik für Neurochirurgie, Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Neurochirurgische Klinik, Universitätsklinikum Gießen und Marburg UKGM, Giessen
  - Klinik für Neurochirurgie, Universitätsmedizin Göttingen, Göttingen
  - Klinik für Neurochirurgie, Klinikum Kassel, Kassel
  - Neurochirurgische Klinik, Universitätsmedizin Mainz, Mainz
  - Neurochirurgische Klinik, Universitätsklinikum Mannheim, Mannheim
  - Dep. of Neurosurgery, Klinikum rechts der Isar der Technischen Universität München, Munich
  - Klinik für Allgemeine Neurologie, Universitätsklinikum Münster, Münster
  - Klinik für Neurochirurgie, Universitätsklinikum Würzburg, Würzburg
- Netherlands (2):
  - Academic Medical Center Amsterdam, Department of Neurology, Amsterdam
  - University Medical Center Utrecht, Department of Neurology, Department of Neurosurgery, Utrecht
- Spain (3):
  - Servicio de Neurocirurgía Bellvitge Hospital, Barcelona
  - Servicio de Neurología, Hospital Universitario La Paz, Madrid
  - Servicios de Neurología, Neurocirugía y Cuidados Intensivos del Hospital Virgen del Rocío, Seville
- Switzerland (4):
  - Dep. of Neurology / Dep. of Neurosurgery, Bern University Hospital, Bern
  - Dep. of Clinical Neuroscience, Service of Neurosurgery, Geneva
  - Dep. Neurosurgery, Ospedale Regionale di Lugano, Lugano
  - Dep. of Neurosurgery, University Hospital Zürich, Zurich

REFERENCES:
- [Derived] Polymeris AA, Lang MF, Hakim A, Butikofer L, Fung C, Beyeler S, Z'Graggen W, Strbian D, Vajkoczy P, Schubert GA, Gruber A, Mielke D, Roelz R, Siepen B, Seiffge DJ, Selim MH, Raabe A, Beck J, Fischer U; SWITCH Study Investigators. Effect of Decompressive Craniectomy According to Location of Deep Intracerebral Hemorrhage: A SWITCH Trial Analysis. Stroke. 2026 Jan;57(1):12-19. doi: 10.1161/STROKEAHA.125.052460. Epub 2025 Oct 17. PMID 41104458
- [Derived] Beck J, Fung C, Strbian D, Butikofer L, Z'Graggen WJ, Lang MF, Beyeler S, Gralla J, Ringel F, Schaller K, Plesnila N, Arnold M, Hacke W, Juni P, Mendelow AD, Stapf C, Al-Shahi Salman R, Bressan J, Lerch S, Hakim A, Martinez-Majander N, Piippo-Karjalainen A, Vajkoczy P, Wolf S, Schubert GA, Hollig A, Veldeman M, Roelz R, Gruber A, Rauch P, Mielke D, Rohde V, Kerz T, Uhl E, Thanasi E, Huttner HB, Kallmunzer B, Jaap Kappelle L, Deinsberger W, Roth C, Lemmens R, Leppert J, Sanmillan JL, Coutinho JM, Hackenberg KAM, Reimann G, Mazighi M, Bassetti CLA, Mattle HP, Raabe A, Fischer U; SWITCH study investigators. Decompressive craniectomy plus best medical treatment versus best medical treatment alone for spontaneous severe deep supratentorial intracerebral haemorrhage: a randomised controlled clinical trial. Lancet. 2024 Jun 1;403(10442):2395-2404. doi: 10.1016/S0140-6736(24)00702-5. Epub 2024 May 15. PMID 38761811
- [Derived] Fischer U, Fung C, Beyeler S, Butikofer L, Z'Graggen W, Ringel F, Gralla J, Schaller K, Plesnila N, Strbian D, Arnold M, Hacke W, Juni P, Mendelow AD, Stapf C, Al-Shahi Salman R, Bressan J, Lerch S, Bassetti CLA, Mattle HP, Raabe A, Beck J. Swiss trial of decompressive craniectomy versus best medical treatment of spontaneous supratentorial intracerebral haemorrhage (SWITCH): an international, multicentre, randomised-controlled, two-arm, assessor-blinded trial. Eur Stroke J. 2024 Sep;9(3):781-788. doi: 10.1177/23969873241231047. Epub 2024 Feb 12. PMID 38347736
- See also: Website of the trial — http://www.switch-trial.ch